CLINICAL TRIAL: NCT07401940
Title: A Multi-Generational Suicide Prevention Program in African American Churches
Brief Title: HAVEN-Connect Youth Suicide Prevention
Acronym: HAVEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Mt. Sinai School of Medicine, New York, New York (Unknown); University of Rochester (Other); American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TBT-0-010-21
Record Dates: First submitted 2025-12-03; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Suicide Prevention
Keywords: suicide prevention; Black youth; church based prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: This study uses a cluster randomized, wait-list design, with youth clustered within churches, and churches randomly assigned to order of implementation within each site. Randomization will occur at the church level since HAVEN is a multi-level, church-based intervention. In each of 3 cohorts, 4-6 churches will be matched as pairs based on location (Harlem/Rochester) and size for a total of 2-3 pairs per cohort (12-18 churches total).
  Youth recruitment and baseline assessments of youth will occur simultaneously with church engagement and the Clergy participating in the Faith Based Curriculum. One church from each matched pair will be randomly assigned to begin HAVEN immediately, and the other to a wait-list condition to receive HAVEN approximately 6 months later. The active phase of evaluating HAVEN will span 6-8 months (8 months for wait-listed churches): a 2 month engagement and church leader curriculum phase, followed by HAVEN=Connect training delivered over 1 month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAVEN Intervention Group (Experimental): Participants receive HAVEN Connect intervention
  Interventions: Behavioral: HAVEN-Connect
- HAVEN Wait List Control Group (Placebo Comparator): On 6-month wait list where they only receive text messages
  Interventions: Behavioral: HAVEN Suicide Prevention

INTERVENTIONS:
Behavioral: HAVEN-Connect — Youth-Connect Program for adolescents/emerging adults and Connect training for adult members is a strength-based network health depression and suicide prevention program. Participants learn together about and model skills to each other to grow and sustain "Four Cores" supportive of mental health and reduced likelihood of vulnerability to suicidal thoughts: (1) Healthy relationships and accountability spanning friendship, community and family relationships (Kinship); (2) Meaning and value in life (Purpose); (3) Informal and formal help-seeking (Guidance); and (4) Activities that give strength and balance emotions (Balance). Modules include self-assessment of strength areas, needs and using Four Cores to manage challenging emotions. Group skill-building activities identify strengths of all members, and members learn how a strong network supports all members' well-being. The training uses active learning including high energy activities and peer-to-peer teaching.
  Arms: HAVEN Intervention Group
Behavioral: HAVEN Suicide Prevention — Connect was developed to extend Sources of Strength, an evidence-based suicide prevention program that trains key opinion leaders to disseminate a model of healthy coping to peers, which has been implemented in over 80 secondary schools in New York State. Connect uses a multiple-session group training to build suicide protection at individual and group levels. The first version, Wingman-Connect was developed for young Air Force personnel in training (20% Black or multiracial).
  Arms: HAVEN Wait List Control Group

SUMMARY:
HAVEN=CONNECT is a comprehensive depression and suicide prevention intervention that is designed to be integrated into predominantly Black churches, a strategically ideal location for mental health intervention for Black youth. HAVEN=CONNECT has three components: (1) Church Community Engagement: an interactive process of introducing the program to key church leaders and stakeholder groups. (2) Faith-Based Curriculum: educational overview for pastors, other ministerial staff and youth lay leaders on how to integrate the program into the church using communication mediums that have cultural and religious relevance in the Black Church context. (3) Youth-Connect Intervention: The goals of this project are to test the impact of HAVEN=CONNECT (HAVEN) on key intervention targets, hypothesized mediators, and build a research-informed implementation strategy for future large-scale testing.

DETAILED DESCRIPTION:
Aim 1: Efficacy. The investigators will implement HAVEN in 12 churches using a cluster randomized waitlist design and enroll 240 adolescents (ages 13-19). The investigators hypothesize that adolescents in HAVEN churches vs. those in wait-listed churches will have decreased depression symptoms (primary outcome) and suicide risk scores at 1-month and 6-month follow-up after the start of the multi-component HAVEN. Suicide risk will be a secondary outcome due to lower expected statistical power to detect impact vs. depression. The investigators also expect HAVEN to decrease other mental health symptoms that are secondary outcomes (e.g., anxiety). The investigators will test for differences by gender, age, and level of depression and suicide risk at baseline.

Aim 2: Mechanisms. The second aim is to test hypothesized mediators of HAVEN impact. It is hypothesized that HAVEN will increase (a) adolescents' positive bonds to peers and adults in their church, perceptions of cohesion, and healthy norms in those networks; (b) emotional and behavior self-regulation, and (c) increased use of mental health services (H1). HAVEN impact on reducing depression and suicide risk will be mediated by those changes (H2).

Aim 3: Implementation. The investigators will identify implementation barriers and facilitators by examining adherence data (i.e., completion of HAVEN steps and clergy/member engagement) and then gathering qualitative data from a subset of 4 churches, 2 identified as implementing HAVEN with high adherence and 2 with lower adherence. This aim involves semi-structured key informant interviews. The investigators will also train church and community members as HAVEN=CONNECT co-trainers, assess their fidelity of training using existing fidelity measures, as part of this aim on identifying strategies for sustaining HAVEN after the end of the grant period and for scalability.

Primary outcome variable for Youth: Suicide risk & depression Secondary outcome variable for Youth: Anxiety Mediators for Youth: mental health service use, emotion regulation skills, stressful life events, adolescent experiences with discrimination, peer networks, help-seeking acceptability, group cohesion, healthy peer norms and behaviors, trusted adult networks, Helpfulness of Adults with emotions, positive communication with parents, demographic information.

Adult mediators: satisfaction with training, retention of skills, intention to use skills in personal life and with youth, adoption of skills, experience engaging youth with skills, and adult peer network.

ELIGIBILITY:
Inclusion Criteria: For churches:

1. 75% of members self-identify as Black or African American,
2. 75% are fluent in English.

Exclusion Criteria for Youth:

1. self-identify as Black/African American,
2. 13-19 years old, are fluent in English

Exclusion Criteria: Churches:

1. 25%+ of members self-identify as non-Black or African American
2. 25%+ are not fluent in English.

Exclusion Criteria for Youth:

1. do not self-identify as Black/African American,
2. are younger than 13 or older than 19.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Kiddie-Computerized Adaptive Testing for Mental Disorders | baseline, 1- and 6-month followup
  Measures depressive symptoms and suicide risk; it asks fewer questions than traditional suicide screeners because it is response adaptive. Instead of fixing the items and allowing the precision of measurement to vary, the authors fix the precision of measurement and allow the items to vary. The K-CAT adaptively selects a small set of items from a large item-bank of 2,120 items, using a 4-point Likert scale (Strongly Agree, Agree, Disagree, Strongly Disagree). The results yield four metrics: 1) a severity score ranging from 0 - 100, with 0 representing the lowest severity, and 100 representing the highest severity. The prompt for each question is: "In the past two weeks..." Sample items include: "I felt worthless" I felt everyone would be better off without me"
  .

SECONDARY OUTCOMES:
Kiddie-Computerized Adaptive Testing for Mental Disorders. | baseline, 1- and 6-month followup
  Description: Measures anxiety symptoms. it asks fewer questions than traditional suicide screeners because it is response adaptive. Instead of fixing the items and allowing the precision of measurement to vary, the authors fix the precision of measurement and allow the items to vary. The K-CAT adaptively selects a small set of items from a large item-bank of 2,120 items, using a 4-point Likert scale (Strongly Agree, Agree, Disagree, Strongly Disagree). The prompt for each question is: "In the past two weeks..."
  Sample items include:
  I worried more than I needed to I felt uneasy much of the time It is hard for me to relax My worries overwhelmed me

OTHER OUTCOMES:
Demographic Questionnaire | baseline
  Measures demographic characteristics of sample (e.g., age, race, gender, gender identity, GPA, etc.). Will be used to describe characteristics of sample and to ascertain if demographic groups respond differently to the prevention program (e.g.., age or gender differences in response to the program.
General Training Satisfaction Questionnaire | baseline (immediately following training
  Adult participants receive a brief set of questions to assess general satisfaction. with the program, n of items = 3. measured on a Likert scale: (0 = not at all - 3 = very much) score range = 0-9 with high scores interpreted as being high training satisfaction.
Retention of Skills Questionnaire | baseline (immediately after training), 3-month follow-up
  Adult participants will receive a brief set of questions to assess perceptions of the training, retention and adoption of training information, and use of concepts in life. n of items = 7. measured on a dichotomous scale: (0 = false, 1 = True) score range = 0-7 with high scores interpreted as high retention of skills learned from the prevention program.
Intention to use HAVEN-Connect Skills Questionnaire | baseline (immediately after training), 3-month follow-up
  Assess perceptions of intention to use the skills learned in the HAVEN prevention program. n of items = 7, measured on a Likert scale: (0 = strongly disagree to 100 = strongly agree). score range = 0-100 (calculate the mean score), with high scores interpreted as having high intentions to use newly acquired skills gained from the training sessions.
Intention to Use Skills with Youth Questionnaire | baseline (immediately after training), 3-month follow-up
  Assess intentions to use newly acquired skills with youth in the future. n of items = 5, measured on a Likert scale: (0 = strongly disagree to 100 = strongly agree). score range = 0-100 (calculate the mean score), with high scores interpreted as having high intentions to use newly acquired skills gained from the training sessions with youth
Adoption of Skills Questionnaire | baseline (immediately after training), 3-month follow-up
  Assess perceptions of the training, retention and adoption of training information, and use of concepts in life. n of items = 5, measured on a Likert scale: (0 = strongly disagree to 100 = strongly agree). score range = 0-100 (calculate the mean score), with high scores interpreted as believing the person will adopt the skills acquired through the program to daily life.
Experience Engaging Youth with Skills Questionnaire | baseline (immediately after training), 3-month follow-up
  Assess use of core concepts in interactions with youth. n of items = 5, measured on a Likert scale: (0 = strongly disagree to 100 = strongly agree). score range = 0-100 (calculate the mean score), with high scores interpreted as having high intentions to actively engage the youth with newly acquired skills gained from the training sessions.
Adult Peer Network Questionnaire | baseline, 3-month follow up
  Adults nominate close friends at church. Asked to name up to 7 adults who serve as a support network for the adults. Range is from 0-7. Higher numbers indicate more peers in peer network.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry D Molock, Ph.D., M.Div., Principal Investigator — George Washington University, Dept of Psychological & Brain Sciences; Sidney Hankerson, MD, MBA, Principal Investigator — Mt. Sinai Icheon School of Medicine - Psychiatry; Peter Wyman, Ph.D., Principal Investigator — University of Rochester Medical Center - Psychiatry
Locations (2):
- United States (2):
  - Mt. Sinai Hospital; Ichon School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
The final data set will include demographic information, outcome data (suicide ideation and attempts, depression, anxiety, PTSD) and possible mediators, including mental health service utilization, peer networks, help-seeking acceptability, peer norms, trusted adult network, etc. Data products will be made available without costs to researchers. User registration is required in order to access or download files. Users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. Registered users will receive user support, information related to errors in the data, future releases, workshops, and publication lists. Data cannot be used for commercial purposes or distributed to third parties
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start Date: June 1, 2029 How long: 2years
Access Criteria: Registered users will have access to: demographic information, outcome data (suicide ideation and attempts, depression, anxiety, PTSD) and possible mediators, including mental health service utilization, peer networks, help-seeking acceptability, peer norms, trusted adult network, etc. Data products will be made available without costs to researchers. Can access data by contacting the PI, who will provide a link to the data.

REFERENCES:
- [Background] Wyman PA, Pisani AR, Brown CH, Yates B, Morgan-DeVelder L, Schmeelk-Cone K, Gibbons RD, Caine ED, Petrova M, Neal-Walden T, Linkh DJ, Matteson A, Simonson J, Pflanz SE. Effect of the Wingman-Connect Upstream Suicide Prevention Program for Air Force Personnel in Training: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2022532. doi: 10.1001/jamanetworkopen.2020.22532. PMID 33084901
- [Background] Molock SD, Matlin S, Barksdale C, Puri R, Lyles J. Developing suicide prevention programs for African American youth in African American churches. Suicide Life Threat Behav. 2008 Jun;38(3):323-33. doi: 10.1521/suli.2008.38.3.323. PMID 18611131
- [Background] Hankerson SH, Weissman MM. Church-based health programs for mental disorders among African Americans: a review. Psychiatr Serv. 2012 Mar;63(3):243-9. doi: 10.1176/appi.ps.201100216. PMID 22388529
- [Background] Gibbons RD, Kupfer DJ, Frank E, Lahey BB, George-Milford BA, Biernesser CL, Porta G, Moore TL, Kim JB, Brent DA. Computerized Adaptive Tests for Rapid and Accurate Assessment of Psychopathology Dimensions in Youth. J Am Acad Child Adolesc Psychiatry. 2020 Nov;59(11):1264-1273. doi: 10.1016/j.jaac.2019.08.009. Epub 2019 Aug 26. PMID 31465832